CLINICAL TRIAL: NCT02153879
Title: Qualitative and Quantitative Characterization of HDL in T2D After Fenofibrate or Niacin Treatment in Spanish Population
Brief Title: Characterization of High Density Lipoprotein (HDL) in Type 2 Diabetes (T2D) After Fenofibrate or Niacin Treatment
Acronym: LOWHDL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Spanish Biomedical Research Centre in Diabetes and Associated Metabolic Disorders (Other)
Responsible Party: Principal Investigator, LUIS MASANA, MD, Professor, Institut Investigacio Sanitaria Pere Virgili
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IISPV-HUSJR-LOWHDL
Record Dates: First submitted 2014-05-26; First posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Type 2 Diabetes Mellitus; Dyslipidemia
Keywords: HDL; Niacin; Fenofibrate; Diabetes; Metabolomics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Diabetes Mellitus | interventions — Fenofibrate; Niacin; MK-0524

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fenofibrate (Experimental): Fenofibrate 145 mg/day for 12 weeks
  Interventions: Drug: Fenofibrate
- Niacin plus Laropiprant (Experimental): Niacin 2g/day plus Laropiprant for 12 weeks
  Interventions: Drug: Niacin plus laropiprant

INTERVENTIONS:
Drug: Fenofibrate — fenofibrate 145/day for 12 weeks
  Other Names: Secalip
  Arms: Fenofibrate
Drug: Niacin plus laropiprant — Niacin 2 g/day plus Laropiprant for 12 weeks
  Other Names: Tredaptive
  Arms: Niacin plus Laropiprant

SUMMARY:
The structural and functional alterations of high density lipoproteins (HDL) levels in type 2 diabetes (T2D) patients linked to hypertriglyceridemia, hyperglycemia, insulin resistance, inflammation and oxidation, play a major role in the increased macrovascular risk in these patients. An impaired function of the adipose tissue (AT) in T2D contributes to low HDL concentrations.

Objectives: 1) Quantitative and qualitative characterisation of HDL subclasses by ultracentrifugation, proteomic and metabolomic techniques. 2) To study the relationship between the HDL subclasses, preβ1 HDL and remnant HDL, and clinical determinants of arteriosclerosis. 3) Functional in vitro studies of the HDL subclasses determined in Objective 1. 4) To study the role of AT determining the low HDL levels. 5) To study the impact of HDL increasing drugs on HDL qualitative changes.

DETAILED DESCRIPTION:
Groups of subjects: a) Diabetic patients with low HDL; b) Non-diabetic patients with low HDL; c) Diabetic patients with normal HDL levels; and d) Non-diabetic patients with normal HDL levels. The studies will be performed after washing out lipid lowering drugs. Intima media thickness (IMT) will be performed in all groups. Main biochemical techniques will be centralised. Isolation and characterisation of HDL subclasses and remnant HDL, as well as a determination and preβ1 HDL will be performed. HDL studies examining HDL proteomic and metabolomic profiles will be performed. Functional studies will determine the effects on the endothelium, inflammation, cholesterol efflux and oxidation according the qualitative changes. These HDL measurements will be repeated in group (a), after they are treated with fibrates or Niacin. HDL metabolism in adipocytes will be extensively studied, and the clinical associations between HDL alterations and plasma AT-derived molecules will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients
* Age from 30 years to 70 years
* HDL not exceeding 50 mg/dl in men or 60 mg/dl in women

Exclusion Criteria:

* to be a smoker
* To be diagnosed with diabetes less than three months before
* To have triglyceride levels above 400 mg/dl
* Glycated hemoglobin higher than 9%
* Albuminuria above 300 mg/mg creatinine
* Chronic kidney disease (eFGR <30 ml/min/1.73 m2)
* Advanced retinopathy
* Neuropathy
* Cardiovascular disease in the last three months
* Chronic liver insufficiency
* Neoplastic disease or any chronic or incapacitating disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
HDL particles size and number assessed by nuclear magnetic resonance (NMR) and reported as nm and micromol/L | Two periods of 12 weeks treatment according to crossing over design
  HDL particles were studied by NMR in T2D patients after treatment with fenofibrate or Niacin

SECONDARY OUTCOMES:
Apolipoprotein A1 (Apo A1), apolipoprotein A2 (Apo A2), paraoxonase (PON) HDL concentration (g/l - mg/l) | Two periods of 12 weeks treatment according to crossing over design
  Apoprotein and antioxidant enzymes composition of HDL were also measured

OTHER OUTCOMES:
Lecithin-cholesterol acyltransferase (LCAT) and cholesteryl ester transfer protein (CETP) activity (AU - pmol/h*μl) and mass (microg/ml) | Two periods of 12 weeks treatment according to crossing over design
  LCAT and CETP mass and activities were measured;

CONTACTS AND LOCATIONS:
Overall Officials: Luis Masana, Professor, Study Director — Institut Investigacio Sanitaria Pere Virgili
Locations (1):
- Hospital Universitari Sant Joan, Reus, Tarragona, Spain

REFERENCES:
- See also: Institut Investigacio Sanitaria Pere Virgili- Pere Virgili Health Research institute — http://www.iispv.cat